CLINICAL TRIAL: NCT03447353
Title: SAFER-SIM: Opiates and Benzodiazepines on Driving
Brief Title: Opiates and Benzodiazepines on Driving
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Timothy L. Brown (Other)
Responsible Party: Sponsor-Investigator, Timothy L. Brown, Associate Research Scientist/Engineer, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 201604731
Record Dates: First submitted 2018-02-07; First posted 2018-02-27 (Actual); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-04

CONDITIONS: Driving Behavior
Keywords: driving; Xanax; Norco; simulation
MeSH Terms: interventions — Alprazolam; Tablets; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- "Sober" or Double Placebo (Experimental): Subject receives two tablets, both containing placebo
  Interventions: Drug: Placebo Oral Tablet
- Active Xanax, Active Norco (Experimental): Subject receives two tablets, one containing Xanax and one containing Norco
  Interventions: Drug: Xanax 1Mg Tablet; Drug: Norco 10Mg-325Mg Tablet
- Active Xanax, Placebo Norco (Experimental): Subject receives two tablets, one containing Xanax and one containing placebo
  Interventions: Drug: Xanax 1Mg Tablet; Drug: Placebo Oral Tablet
- Placebo Xanax, Active Norco (Experimental): Subject receives two tablets, one containing Norco and one containing placebo
  Interventions: Drug: Norco 10Mg-325Mg Tablet; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Xanax 1Mg Tablet — Single dose on two of four visits, one in conjunction with 1 tab of 10mg/325mg Norco
  Other Names: Alprazolam
  Arms: Active Xanax, Active Norco; Active Xanax, Placebo Norco
Drug: Norco 10Mg-325Mg Tablet — Single dose on two of the four study visits, one in conjunction with 1mg alprazolam
  Other Names: hydrocodone/acetaminophen
  Arms: Active Xanax, Active Norco; Placebo Xanax, Active Norco
Drug: Placebo Oral Tablet — Single dose on two of the four study visits, double dose on one of the four study visits
  Arms: "Sober" or Double Placebo; Active Xanax, Placebo Norco; Placebo Xanax, Active Norco

SUMMARY:
The aim of this research is to assess drug effects (Xanax and Norco) on driving performance. Researchers will use the Alertness Memory Profiler (AMP) application to compare results to previous related studies.

This study continues a line of research designed to characterize the effects of common recreationally used prescription and illicit drugs with well known stimulant and sedating effects and their relationship to results from the Alertness Memory Profiler (AMP) that included a set of vigilance and memory tasks.

DETAILED DESCRIPTION:
This study uses EEG, EKG, computerized assessment, blood sampling, and driving simulation.

Individuals recruited will be normal, healthy individuals not currently taking the study drugs. The study will involve five visits, a screening visit as well as four dosing visits. The dosing visits will have a clean (double placebo) and three drugged visits (Xanax and Norco placebo, Xanax placebo and Norco, Xanax and Norco). The screening visit will last about two hours and will include drug and pregnancy testing as well as screening for physical/psychological health. Each of the dosing visits will last approximately five to six hours and will include sleep and food intake surveys, being dosed with study drugs or placebos, AMP assessments, a simulator drive, and wellness surveys. There will also be 4 mL blood sampling before dosing, before driving, and after driving.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women, based on medical and psychological evaluation
* Currently valid unrestricted (except for vision correction) US driver's license
* Licensed driver for at least the past two years
* Drove at least 5000 miles in the past year, by self-report
* Live within a 60 mile radius of NADS
* Available for five study sessions, with one being approximately 2 hours and four being approximately 5-6 hours
* Peripheral veins suitable for repeated venipuncture
* Systolic blood pressure within a clinically normal range (120 ± 30 mmHg) and diastolic blood pressure of 80 ± 20 mmHg
* Good command of written and spoken English
* Female subjects with reproductive potential must agree to use (and/or have their partner use) one (1) acceptable method of birth control beginning at the screening visit throughout the study (including intervals between treatment periods/panels) and until 2 weeks after the last dose of study drug in the last treatment period. Acceptable methods of birth control include the following: intrauterine device (IUD-with or without local hormone release), diaphragm, spermicides, cervical cap, contraceptive sponge, oral contraceptives or condoms. Abstinence is an alternative lifestyle and subjects practicing abstinence may be included in the study.

Exclusion Criteria:

* Requires any special equipment to help drive, such as pedal extensions, hand brake or throttle, spinner wheel knobs, or other non-standard equipment
* Presence of any clinically significant illness, as detected by history, physical examination, and/or laboratory tests, that might influence driving performance (e.g., seizures, sleep apnea, narcolepsy, vertigo, chronic fatigue syndrome) or put the subject at increased risk of adverse events (e.g., cardiac arrhythmia, hypertension)
* If female, pregnant or nursing
* Currently taking drugs that are contraindicated for use with study drugs
* Significant history of motion sickness or demonstrates significant simulator sickness during practice drives at screening (SSQ). Subjects must have scores below the following values on the SSQ: Nausea < 21, Oculomotor <32, Disorientation < 15, and Total Score < 32.
* History of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the subject from study participation
* Prior participation in a driver impairment or distraction-related research study conducted at NADS that uses the same base drive

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Brown, Ph.D., Principal Investigator — National Advanced Driving Simulator at the University of Iowa
Locations (1):
- National Advanced Driving Simulator, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Individuals who completed the study completed all four arms of the study and the data is aggregated. Subjects who did not complete the study may have completed one arm and their data is not included in the analysis. There was a screening visit and four study visits where the subject arrived at the National Advanced Driving Simulator. At each study visit, subjects received one of the following four dosing regimens: double placebo or "Sober"; active Xanax with active Norco, active Xanax and placebo Norco, and placebo Xanax and active Norco.
Period: Overall Study
Arm/Group | Overall Study
Started | 18
Completed | 8
Not Completed | 10
Not completed — Failure at Screening Visit | 2
Not completed — Lost to Follow-up | 4
Not completed — Scheduling Conflicts | 3
Not completed — Withdrew - Nausea Study V1, Sim Drive | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to receive all interventions.
  "Sober" or Double Placebo: Participant receives two tablets, both containing placebo.
  Active Xanax, Active Norco: Participant receives two tablets, one containing Xanax and one containing Norco Active Xanax, Placebo Norco: Participant receives two tablets, one containing Xanax and one containing placebo Placebo Xanax, Active Norco: Participant receives two tablets, one containing Norco and one containing placebo
  Placebo Oral Tablet: Single dose on two of the four study visits, double dose on one of the four study visits Xanax 1Mg Tablet: Single dose on two of four visits, one in conjunction with 1 tab of 10mg/325mg Norco Norco 10Mg-325Mg Tablet: Single dose on two of the four study visits, one in conjunction with 1mg alprazolam
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: SDLP
Description: Standard Deviation of Lane Position
  Standard deviation of lane position was analyzed using the SAS GLM function to identify changes in driver performance. Values represents means across the driving environments studied.
Time Frame: over course of each simulator drive, approximately 35 minutes per visit
Population: For the purposes of analysis, the individual interventions are broken down to observe differences. Each of the 8 participants experienced the 4 interventions, in varying order, so each intervention will have 8 overall participants analyzed.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | "Sober" or Double Placebo | Active Xanax, Active Norco | Active Xanax, Placebo Norco | Placebo Xanax, Active Norco
Number analyzed (Participants) | 8 | 8 | 8 | 8
centimeters | 35.2 (11.1) | 49.8 (21.0) | 50.0 (25.3) | 33.5 (9.5)

2. Secondary Outcome: Lane Departures
Description: Total number of lane departures per drive
  The total number of lane departures across the drive were analyzed using the SAS GLM procedure.
Time Frame: over course of each simulator drive, approximately 35 minutes per visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: count
Arm/Group | "Sober" or Double Placebo | Active Xanax, Active Norco | Active Xanax, Placebo Norco | Placebo Xanax, Active Norco
Number analyzed (Participants) | 8 | 8 | 8 | 8
count | 23.8 (9.0) | 72.0 (38.2) | 64.4 (29.4) | 22.3 (9.5)

ADVERSE EVENTS:
Groups:
- "Sober" or Double Placebo: Participant receives two tablets, both containing placebo.
- Active Xanax, Active Norco: Participant receives two tablets, one containing Xanax and one containing Norco
  Xanax 1Mg Tablet: Single dose on two of four visits, one in conjunction with 1 tab of 10mg/325mg Norco Norco 10Mg-325Mg Tablet: Single dose on two of the four study visits, one in conjunction with 1mg alprazolam
- Active Xanax, Placebo Norco: Participant receives two tablets, one containing Xanax and one containing placebo
  Xanax 1Mg Tablet: Single dose on two of four visits, one in conjunction with 1 tab of 10mg/325mg Norco
- Placebo Xanax, Active Norco: Participant receives two tablets, one containing Norco and one containing placebo
  Norco 10Mg-325Mg Tablet: Single dose on two of the four study visits, one in conjunction with 1mg alprazolam
Arm/Group | "Sober" or Double Placebo | Active Xanax, Active Norco | Active Xanax, Placebo Norco | Placebo Xanax, Active Norco
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No